CLINICAL TRIAL: NCT03048903
Title: The Effect of Rhubarb on Sepsis and Post-traumatic Gastrointestinal Function
Brief Title: The Effect of Rhubarb on Sepsis and Post-traumatic Gastrointestinal Function Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHEN De-chang (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Sponsor-Investigator, CHEN De-chang, Director, Head of Intensive care unit, Principal Investigator, Clinical Professor, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHCZHJJ01; SHCZHJJ01-CDC (Registry Identifier: CHEN De-chang)
Record Dates: First submitted 2017-01-19; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Sepsis
Keywords: Gastrointestinal dysfunction; sepsis; trauma
MeSH Terms: conditions — Sepsis; Wounds and Injuries | interventions — Starch

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into two groups ,using rheum palmatum or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rheum Palmatum Root (Experimental): Rheum Palmatum Root is commercially certified rhubarb(Rheum palmatum ,Sichuan origin, provided by the pharmacy of my hospital)
  Interventions: Drug: Rheum Palmatum Root
- Starch Corn (Placebo Comparator): Medical Starch is harmless to people
  Interventions: Drug: Starch Corn

INTERVENTIONS:
Drug: Rheum Palmatum Root — Rhubarb is commercially certified rhubarb(Rheum palmatum , Sichuan origin, provided by the pharmacy of my hospital), ground into a powder, over 80 mesh steel mesh.The dose is 6g in the first 2 days, 3 times / day, oral or nasal feeding,two days later the dose is reduced to 3g, three times / day, oral or nasal feeding.
  Other Names: Chinese Rhubarb Root
  Arms: Rheum Palmatum Root
Drug: Starch Corn — Starch Corn is harmless to people .The use dosage is same as Rheum Palmaturn Root.The dose is 6g in the first 2 days, 3 times / day, oral or nasal feeding,two days later the dose is reduced to 3g, three times / day, oral or nasal feeding.
  Other Names: Medical Starch
  Arms: Starch Corn

SUMMARY:
Random grouping by computer, divided into two groups, a group of rhubarb treatment group, another group for the placebo group.

DETAILED DESCRIPTION:
Patients were randomly divided into two groups, using rhubarb powder or placebo. Rhubarb is commercially certified rhubarb(Rheum palmatum, Sichuan origin, provided by the pharmacy of my hospital), ground into a powder, over 80 mesh steel mesh, Two days before 6g, three times / day, oral or nasal feeding, two days later reduced to 3g, three times / day, oral or nasal feeding; Another group of patients taking placebo, with the same dose of Rhubarb; The overall course of the two drugs was a week.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-65 year old;
2. Diagnosis: sepsis with gastrointestinal dysfunction (II-III grade AGI); gastrointestinal dysfunction after trauma (II-III AGI);
3. Complete gastrointestinal tract anatomic structure（including the ileum and colon stoma）

Exclusion Criteria:

1. Hemodynamic instability;
2. Underlying diseases: cardiac function III~IV, chronic liver dysfunction Child-Pugh score >9 points;
3. Less than 5 days after surgery for stomach and small intestine，less than 7 days after Colonic surgery, Postoperative gastrointestinal leakage;
4. Abdominal Compartment Syndrome;
5. mechanical ileus
6. active gastrointestinal hemorrhage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
The remission rate of gastrointestinal dysfunction | 2 weeks
  The rate of patients who can tolerate 1000Kcal whole protein enteral nutrition in all subjects

SECONDARY OUTCOMES:
The ratios of L/M in human urine samples | 7 days
  The ratios oflactulose / mannitol in human urine samples
citrulline | 7 days
  The contents of citrulline in human serum samples
D- lactic acid | 7 days
  The contents of citrulline in human serum samples

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai ChangZheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kubica P, Kot-Wasik A, Wasik A, Namiesnik J, Landowski P. Modern approach for determination of lactulose, mannitol and sucrose in human urine using HPLC-MS/MS for the studies of intestinal and upper digestive tract permeability. J Chromatogr B Analyt Technol Biomed Life Sci. 2012 Oct 15;907:34-40. doi: 10.1016/j.jchromb.2012.08.031. Epub 2012 Sep 4. PMID 22985725